CLINICAL TRIAL: NCT05256784
Title: Mountain Food, as a Natural Probiotic. Evidence From Central and Eastern European Nutrition and Behavior
Brief Title: Mountain Food and Natural Probiotic in Nutrition
Status: Completed | Type: Observational
Sponsor: Zealandina Agency (Other)
Responsible Party: Sponsor
Other Study IDs: Zealandina
Record Dates: First submitted 2022-02-02; First posted 2022-02-25 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-03

CONDITIONS: Immune Deficiency
MeSH Terms: conditions — Immunologic Deficiency Syndromes

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Probiotic 1: Four members of an extended family: 1 white man of 71 years, 1 white woman of 75 years, 1 white man of 44 years, and 1 white woman of 44 years.
  Interventions: Combination Product: Natural probiotics

INTERVENTIONS:
Combination Product: Natural probiotics — Two of the group members use daily Allium Sativum - garlic, one use Natural honey, and 1 Yogurt. It is verifying the immunity of the organism after 40 days of using natural probitotics.

SUMMARY:
Background/Objectives: The research discusses the importance of mountain foods/products and services in the context of healthier nutrition and behavior with the application to agribusiness. The purpose of the research is to highlight the necessity of human behavior in consuming mountain products as natural probiotics.

Subjects/methods: As evidence, the research analyses mountain food and the associated entrepreneurship for Austria and other Central and Eastern European countries (foods/products and services), especially from the mountain area. The authors realized experimental research regarding representative mountain food from Central and Eastern European areas and used the Eurostat database. Data has been taken from Eurostat and processed in Excel and SPSS, using similar models of analysis from published research. Experimental analysis has been realized by the authors and collected from different recognized sources.

DETAILED DESCRIPTION:
The study is focused on performing qualitative research for natural yogurt (animal resource), Allium sativum - garlic (plant resource), experimental analysis for natural honey (apicultural resource), namely honey-dew (manna) which is a mountain product from Maramureș, a region of Romania, and polyflora honey (Tilia - linden with mountain flowers) which is a hilly product from Moldova, a region of Romania, and clinical study on all the mountain products reminded before.

After this study, it will be a comparative study of consumer behavior of mountain products from Central and Eastern European countries and Central and Southern states from the USA.

This study is referring strictly to Central and Eastern European countries, especially Romania (but a country like Romania is representative of the other studied countries). The members of the family which will participate in the study will consume the probiotics reminded before. The family members, participants in the study, are consuming daily natural honey (one member of the family), yogurt (one member of the family), and garlic (two of them). After every 40 days, it will be verified, through laboratory analysis, the level of organism immunity. The analysis will be realized in Synevo Romania. It will be verified Biochemistry: Serum Calcium, Serum Magnesium, Serum Iron (Sideremia); Immunochemistry: Vitamin B12, Serum Folate, Vitamin 25-OH; Hematology: Leukocyte blood count with Hb, Ht, and indices (Leukocyte count, Erythrocyte count, Hemoglobin, Hematocrit, Mean erythrocyte volume, Mean erythrocyte hemoglobin, Mean Hb / erythrocyte concentration, Erythrocyte distribution width, Platelet count, L platelet count platelet distribution, Neutrophil, Lymphocyte, Monocyte, Eosinophil, Basophil); Zinc in the blood.

It will be verified if properly used mountain animal and vegetal resources can become powerful fighters as natural probiotics against various diseases, or to prevent different immunity problems.

Fermented natural dairy products are an extremely important component in the diet of the CEE population, especially for the rural population. Dairy products are often used as natural probiotics, especially within CEE countries. And, the most used mountain product is yogurt (or derivate products similar wit it, such as kefir, ayran, and so on). Within CEE countries, the most important species isolated from lactic bacteria fermented or raw products of dairy origin, are Lactococcus lactis, Leuconostoc sp., and Enterococcus sp. Probiotic dairy products have been analyzed and shown that in addition to nutritional benefits, they positively influence the physiology of the human body. The best-known dairy products are ice cream, cheese, yogurt, milk enriched with strains of Acidophilus and Bifidus, ayran, kefir, and kumis. Dairy drinks (fermented or unfermented) are considered foods that provide probiotics. In the fermentation process, lactic, acetic, and citric acid are naturally obtained, acids that are frequently used in the food industry to improve the organoleptic qualities of several products intended for consumption. The father of the paradigm according to which yogurt is one of the most powerful probiotics, especially for the digestive system, was Elie Metchnikoff, Nobel Laureate for Medicine. He postulated in the famous public presentation "Old Age", held at the Society of French Agriculturalists in Paris on June 8, 1904, that the dependence between lactic acid bacteria and food makes it possible to apply methods to modify the intestinal flora by replacing bad bacteria with beneficial ones. He suggested that yogurt bacteria prevent and annihilate intestinal bacterial infections and hypothesize that regular yogurt consumption prolongs life. Lactic acid bacteria produce microbial metabolism, and the effect is a decrease in intestinal pH, which stops the proliferation of various proteolytic bacterial species. In this way, Metchnikoff kicks off the popularization of yogurt in Europe as a functional food with health benefits.

Regarding plant resources, CEE countries are specialized in using different plants as natural probiotics. But, the most used plant resource is Allium sativum (garlic). Garlic consumption, as a natural probiotic, is just as old in the CEE as in many other countries around the world. Garlic is listed in the Dietary Guide for Americans 2015-2020. Garlic intake variants (capsules, aqueous extract, old alcoholic extract, etc.) are not very popular in the CEE, the preference being clear for the raw version.

The experimental analysis of the study, realized by the authors in accordance with Romanian Research-Development National Institute for Apiculture - Bulletin analysis 39/29.01.2021, show that both types of natural honey have the same diastase index, meaning 29.4±0.18 unities on Goethe; mountain honey has sucrose (β-D-Fructofuranosyl α-D-glucopyranoside) of 2.41±0.43 %, g/g, while hilly products have 2.19±0.39 %, g/g; reducing sugar is in percent of 76.18±3.40 %, g/g and to the other of 75.67±3.37 %, g/g; 5-Hydroxymethylfurfural has a value of 0.10±0.01 mg/100g of honey for the mountain product and 0.19±0.03; mg/100g of honey for the hilly product; mountain honey has a superior PH value of 3.00±0.46 milliliters Sodium hydroxide solutions 1N/100 g of honey and the other of 2.80±0.43 milliliters Sodium hydroxide solutions 1N/100 g of honey; moisture contents has a percentage of 17.20±0.24 %, g/g for the mountain product and of 16.80±0.24 %, g/g for the other type of honey; pollen analysis present percentages of 98% of manna and 2% of mountain polyflora for the mountain product and of 95% of linden and 5% of manna for the other type of mountain; electrical conductivity present a value of 0.55 mS/cm, while ashes are in the value of 0,21±0,02 %, g/g (mountain product) and 0,44±0,03 %, g/g (hilly product); fructose (3S,4R,5R)-1,3,4,5,6-Pentahydroxyhexan-2-one) present a percentage of 41.06 %, g/g (mountain honey) and 40.10 %, g/g (hilly honey) and glucose (2R,3S,4R,5R)-2,3,4,5,6-Pentahydroxyhexanal) a percentage of 35.12 %, g/g (mountain product) and 35.57 %, g/g (hilly product). The physicochemical analysis shows that mountain honey has more qualitative values than hilly honey. Honey-dew (manna) contains minerals (calcium, magnesium, iron, potassium, phosphorus, selenium), antioxidants, organic acids, bioflavonoids, vitamins (especially C and group B), inhibin (strong bactericide), and enzymes. Minerals, proteins, and some acids are found in amounts five to ten times higher in mountain honey than in hilly honey.

It has been verified if properly used mountain animals and vegetal resources (as natural probiotics) can prevent or fight for human immunity.

Regarding Yogurt consumption, the influence on human immunity presents considerable values for magnesium, vitamin D, leukocyte, mean corpuscular hemoglobin, average hemoglobin/erythrocyte concentration, lymphocyte, monocyte, eosinophilic, basophil, and zinc. Different studies confirm the positive influence of yogurt consumption on immunity, as Yang et al. (2022), Ravindran et al. (2022), Kim et al. (2020), Gasparri et al. (2019), Meydani (2000), Leonard (2018), Jafari et al. (2016), Ajibola et al. (2012), Asemi et al. (2012). Allium sativum (garlic) influence positively the immunity of the organism, modifying the values of vitamin D, erythrocyte distribution width, platelets, and platelet distribution width, neutrophil, monocyte, and zinc. The influence of garlic on immunity is confirmed by numerous studies, such as Bandyopadhyay et al. (2021), Singh et al. (2021), Eor et al. (2020), Lee et al. (2020), Champagne et al. (2018), Divya et. al (2017), Percival (2016), Gholipour Kanani et al. (2014), Ried et al. (2014), Hamlaoui-Gasmi et al. (2012), Samson et al. (2012), Mukherjee et al. (2006), Hodge et al. (2002), Oluwole (2001), etc. Natural honey, especially manna honey, is considered to be one of the most powerful fighters of human immunity. According to our clinical analysis mountain honey has a positive effect on the adjustment of calcium, magnesium, vitamin B12, folates, vitamin D, mean corpuscular hemoglobin (MCH), Average Hgb / erythrocyte concentration, erythrocyte distribution width, platelets, lymphocyte, monocyte and eosinophilic. Complex research, clinical and experimental, sustain the importance of natural honey in immunodeficiency, studies as Attia et al. (2022), Bakour et al. (2022), Martínez-Puc et al. (2022), Ismail et al. (2022), Abdulrhman (2018), Sell et al. (2012), Ahmed et al. (2011), Al-Waili (2003), Kitzes (1943).

ELIGIBILITY:
Inclusion Criteria:

* members of the same extended family

Exclusion Criteria:

* outside of the family

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Members of the same family, white men, and women from 44 to 75 years, have minor problems with immunity in the COVID-19 context.
Sampling Method: Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2022-01-26 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Laboratory blood tests 1 | September 2021 - April 2022
  Serum Calcium
Laboratory blood tests 2 | September 2021 - April 2022
  Serum Magnesium
Laboratory blood tests 3 | September 2021 - April 2022
  Serum Iron (Sideremia)
Laboratory blood tests 4 | September 2021 - April 2022
  Vitamin B12
Laboratory blood tests 5 | September 2021 - April 2022
  Serum Folate
Laboratory blood tests 6 | September 2021 - April 2022
  Vitamin 25-OH
Laboratory blood tests 7 | September 2021 - April 2022
  Leukocyte count
Laboratory blood tests 8 | September 2021 - April 2022
  Erythrocyte count
Laboratory blood tests 9 | September 2021 - April 2022
  Hemoglobin
Laboratory blood tests 10 | September 2021 - April 2022
  Hematocrit
Laboratory blood tests 11 | September 2021 - April 2022
  Mean erythrocyte volume
Laboratory blood tests 12 | September 2021 - April 2022
  Mean erythrocyte hemoglobin
Laboratory blood tests 13 | September 2021 - April 2022
  Mean Hb / erythrocyte concentration
Laboratory blood tests 14 | September 2021 - April 2022
  Erythrocyte distribution width
Laboratory blood tests 15 | September 2021 - April 2022
  Platelet count
Laboratory blood tests 16 | September 2021 - April 2022
  L platelet count platelet distribution
Laboratory blood tests 17 | September 2021 - April 2022
  Neutrophil
Laboratory blood tests 18 | September 2021 - April 2022
  Lymphocyte
Laboratory blood tests 19 | September 2021 - April 2022
  Monocyte
Laboratory blood tests 20 | September 2021 - April 2022
  Eosinophil
Laboratory blood tests 21 | September 2021 - April 2022
  Basophil
Laboratory blood tests 22 | September 2021 - April 2022
  Zinc in the blood

CONTACTS AND LOCATIONS:
Overall Officials: Brindusa Covaci, Ph.D., Study Director — Zealandina Agency & Centre for Mountain Economy; Mihai Covaci, Ph.D., Principal Investigator — Zealandina Agency & Hyperion University
Locations (1):
- Zealandina Agency, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The family members, participants in the study, have consumed daily natural honey, yogurt, and garlic. After every 40 days, it has been verified, through laboratory analysis, the level of organism immunity. The analysis has been realized in different laboratories in Romania. It has been verified Biochemistry: Serum Calcium, Serum Magnesium, Serum Iron; Immunochemistry: Vitamin B12, Serum Folate, Vitamin 25-OH; Hematology: Leukocyte blood count with Hb, Ht, and indices (Leukocyte count, Erythrocyte count, Hemoglobin, Hematocrit, Mean erythrocyte volume, Mean erythrocyte hemoglobin, Mean Hb / erythrocyte concentration, Erythrocyte distribution width, Platelet count, Platelet distribution, Neutrophil, Lymphocyte, Monocyte, Eosinophil, Basophil); Zinc in the blood.
  Clinical studies and survival analysis realized for the research show that the immunity of the tested subjects has been improved during mountain products consumption (see detailed description).
Supporting Information: Study Protocol, CSR
Time Frame: September 2021 - April 2022
Access Criteria: Anyone
URL: http://zealanadinaagency.iwopop.com/